CLINICAL TRIAL: NCT04413422
Title: Upper Esophageal Sphincter Pressure Variation During Anesthesia Induction
Brief Title: Study on General Population of the Effect on Airway Protection of Drugs Used During Induction of General Anesthesia
Status: Completed | Type: Observational
Sponsor: Hospital San Carlos, Madrid (Other)
Responsible Party: Principal Investigator, Elena Sanz Sanjosé, Principal Investigator, Hospital San Carlos, Madrid
Other Study IDs: 16/215-O
Record Dates: First submitted 2020-05-18; First posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Aspiration
Keywords: upper esophageal sphincter; propofol; etomidate; thiopental; high resolution manometry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (3):
- propofol: Those patients planned for general surgery, who received propofol as an induction agent for general anesthesia.
  Interventions: Drug: type of hypnotic used for induction of general anesthesia
- etomidate: Those patients planned for general surgery, who received etomidate as an induction agent for general anesthesia.
  Interventions: Drug: type of hypnotic used for induction of general anesthesia
- thiopental: Those patients planned for general surgery, who received thiopental as an induction agent for general anesthesia.
  Interventions: Drug: type of hypnotic used for induction of general anesthesia

INTERVENTIONS:
Drug: type of hypnotic used for induction of general anesthesia

SUMMARY:
Upper esophageal sphincter is a high pressure zone of the pharynx and protects airway from aspiration of esophageal or gastric contents. Existing literature concludes that many of the drugs employed to induce general anesthesia descend that pressure. However, most participants of those studies were under 64 years old and were given sedatives or local anesthetics to ease the esophageal measurements which can interfere with the results obtained. The hypothesis was to confirm the hypnotics effects on upper esophageal sphincter with the aim to find out which of them could be a better choice in order to reduce airway aspiration risk during induction of anesthesia, specially during emergency surgery, when a empty stomach is not guaranteed. Twenty patients who were planned for general surgery were studied: 12 men and 8 women, aged 39 to 84 years old. The effect of three commonly used hypnotics was tested: propofol, etomidate, and thiopental. Written informed consent was explained to all participants who freely signed it after having understood and accepted it. After 6-8 hours fast, patients were monitored with entropy (which gives information about patients´ level of consciousness), electrocardiogram, pulse oximetry (measures blood oxygen), and sphingomanometry (measures blood pressure). Registry of upper esophageal sphincter pressure was obtained through solid state high resolution manometry. A lubricated manometric probe was introduced through the nostril to locate it from the pharynx to the stomach using no sedation. After 1 minute to make the patient feel more comfortable, the induction of anesthesia took place employing one of the three drugs for this purpose mentioned above. Comparison of upper esophageal sphincter pressures before and after the hypnotic administration, should give information about which of the three hypnotics, if any, would not led to an unprotected airway and so at increased risk of aspiration.

DETAILED DESCRIPTION:
BACKGROUND

Upper esophageal sphincter is a high pressure zone, behind the cricoid cartilage, which protects airway from aspiration. It consists on striated muscle fibers distributed in two zones: rapid twich oblique fibers correspondent to tyropharyngeal muscle and rapid but mostly slow twich horizontal fibers belonging to cricopharyngeal muscle. This permits sphincter maintain a constant basal tone but, at the same time, respond quickly to reflexes (1).

Upper esophageal sphincter pressure is distributed asymmetrically being greater anteroposteriorly than laterally. Peak anterior pressure is located more cranially than peak posterior pressure (2).

This makes manometric measurements difficult and some unreliable, unless high resolution manometry is used. Upper esophageal sphincter pressure is labile: it decreases with age and deterioration of the level of consciousness; while increases with stress, anxiety, inspiration and phonation. Patients referring dysphagia or gastroesophageal reflux may present altered manometric measurements (3).

Upper esophageal sphincter has a dynamic function, taking part during burps, in deglutition, and airway reflexes such as: esophagus-sphincter reflex, glottic- pharynx reflex and coughing ( 3).

Studies using propofol and sevoflurane at subhypnotic concentrations have shown a decrease in upper esophageal sphincter pressure, as well as pharynx descoordination (4). Midazolam at sedative doses was implicated in lowering upper esophageal sphincter pressure. Vanner et al made an anesthesia induction using midazolam, thiopental or ketamine, concluding that, except for the last one, all drugs caused a decrease in upper esophageal sphincter pressure. In another study of the same working group, inhalational anesthesia using protoxide and halothane was compared to intravenous anesthesia with thiopental. Upper esophageal sphincter pressure only descended under thiopental (5,6).

Since aspiration depends not only on upper esophageal sphincter but also on lower esophageal sphincter and barrier pressure, it is important to know how drugs affect them: Thiopental, opiates, dexmedetomidine and propofol may diminish lower esophageal sphincter tone (7).

Thörn K. et al studied the effect of sevoflurane on lower esophageal sphincter pressure and barrier pressure, objecting a statistically significant descend in both of them (8).

Some studies do not find an implication of propofol in lowering upper esophageal pressure (9).

Propofol, etomidate, and thiopental effect on upper esophageal sphincter pressure was evaluated in this study. All of them potentiate the inhibitory effect of GABA (gamma-amino-butiric acid) neurotransmisor; etomidate and thiopental also depress ascending activating reticular system. To measure how they affect level of consciousness, entropy, a parameter obtained from electroencephalic signal registration, has been used. Specifically, State Entropy (SE) was used, which computes over the frequency range of 0,8 to 32 Hz. Entropy monitoring has been validated using different hypnotics, being compared to other types of EEG records , as Bispectral Index (BIS) (10).

General anesthesia procedure for patients undergoing urgent surgery is usually done following a "rapid sequence technique". In addition to the possibility of existing full stomach, airway protection mechanisms may be altered during induction. That is why, finding a hypnotic, not to affect or in a lesser manner, upper esophageal sphincter, would be of interest.

PATIENTS AND METHODS Duly approved by the ethics comitee of Clínico San Carlos Hospital of Madrid in their meeting on the 8th of june of 2016 (act 6.1/16) the study was carried out between january of 2017 and july of 2019. 43 patients to be going under general anesthesia for programmed surgery were included, of which: 15 rejected taking part of the study; 3 did not pass dysphagia or reflux tests; 5 patients were lost due to different causes (2 did not tolerate the probe; in 2 cases the protocol failed; in 1 case there was a bias in manometric measurements).

Finally, the study was reduced to 20 patients: 12 men and 8 women, aged between 39 and 84 years old; mean age was 65,05 (13,13). In reference to anesthetic risk, 15% of patients were ASA I, 55% ASA II, and 30% were ASA III. Mean (sd) Body Mass Index was 26.70 (4.24) kg/m2.

Written informed consent was explained to all patients who freely signed it after having understood and accepted it. Patients were distributed randomly in 3 groups depending on the hypnotics they were receiving. During the progress of the investigation, given the difficulties to find people who wanted to participate in the study, the comparative was reduced to only 2 groups: propofol and etomidate. This explains the definitive distribution: 8 patients in propofol group; 9 in etomidate group; 3 in thiopental group.

Two anesthesiologists worked as research collaborators during each case. One of them was in charge of proceeding with the induction as the protocol dictated, and another research collaborator was exclusivelly dedicated to the informatic registry of all the parameters, recording all together for each patient in a single archive corresponding to each participant. A doctor specialized in gastroenterology, expert on manometry, was responsible for introducing the manometric probe and making the consequent measurements, synchronizing his work with that of the other two research collaborators mentioned above.

Once all data had been recorded, the main investigator, who ignored which medication had been given to each patient, gathered all the information together. Each hypnotic had been assigned to a different color so each patient was associated to a color and a number. In this way, any influence on the interpretation of the results was avoided.

The protocol was as follows: After 6-8 hours fast, patients were monitored with entropy (spectral entropy monitoring module, Healthcare Technologies ®), electrocardiogram, pulse oximetry, and sphingomanometry (hemodynamic and respiratory monitoring module for S/5Avance®, General Electric). A lubricated manometric probe was introduced through the nostril to locate it from the pharynx to the stomach using no sedation. After 1 minute to permit the patient get used to the probe and be calm. while receiving oxygen at 10 lpm through a face mask., an initial (basal) manometric measure was noted. In this moment, the hypnotic was administered during 30 s. (to emulate rapid-sequence induction) at the following doses: 2 mg/kg for propofol, 0.4 mg/kg for etomidate or 4 mg/kg for thiopental. Afterwards, once entropy reached a value of 60, a second measure of upper esophageal sphincter pressure was noted. In case entropy did not fall to 60 or less, it was waited the necessary time for the hypnotic to make its effect on level of consciousness (clinical signs such as loss of response, loss of eyelid reflex, absence of sympathetic system activation such as tachycardia or hypertension were indications of the patient´s state of consciousness in those cases). All measurements except for manometry were recorded with an interval of 1 second through Datex-OhmedaTM S/5 Collect® and data were collected in an excel chart. Later, it is all analized combining manometric, entropy, hemodynamic and respiratory measurements. In case of oxygen saturation values of 93% or less or mean arterial pressure descending 20% or more from basal, the record was stopped.

Statistical analysis Quantitative variables are described as median and interquartile range due to their no normal distribution in this study. Due to the small size of the sample no parametric tests are used. The study of the change that hypnotics cause on quantitative variables is carried out through Wilcoxon test. Analizing differences between groups, thiopental group is not taken into account given the small size of it. As a result, statistical tests used to compare variables between different hypnotics do not include thiopental group. Homogeneity of propofol and etomidate group is checked out through Mann- Whitney or Chi squared test depending on the type of variable under study, quantitative or cualitative, respectively. The study of parameters of interest (upper esophageal sphincter pressure; entropy) drop is done through the percentage of change they experiment after the hypnotic has been administered. The relationship of these two variables between both groups of hypnotics is analyzed by Mann- Whitney test. Level of significance is considered of 5%. Statistical software used was IBM SPSS Statistics v21.

ELIGIBILITY:
Inclusion Criteria:

Candidates ought to comply with all these conditions:

* Had been classified by an anesthesiologist (not participating in the study) , at the preanesthetic consult as I, II or III class from the ASA (American Society of Anesthesiologists) classification in reference to his/her anesthetic risk.
* Patients of any gender.
* Patients aged 35 to 85 years old.
* Candidates to planned general surgery to be given general anesthesia.
* Be correctly informed through orally and in writing about the study.
* Voluntary acceptance to participate in the study, voluntary signing the informed consent , which could be revoked at any time through the study.
* Not presenting any of the exclusion criteria.

Exclusion Criteria:

* Presenting known allergy or hypersensitivity to any of the drugs to be potentially administered.
* Pregnancy.
* Psychiatric history or being on treatment with psychotropic drugs.
* Being on treatment with any of these drugs (which can cause alterations in esophageal motility): prokinetics, sedatives, calcium channel antagonists, nitrates, anticholinergics, tricyclic antidepressants, teophyline.
* Having had esophageal surgery.
* Those who, from an anesthetic or medical point of view could present complications during the process. For example: difficult airway or problems with ventilation.
* Renal or hepatic alteration which may interfere with hypnotics pharmacokinetics.
* Renounce to sign informed consent, therefore not authorizing to participate in the study.
* Not presenting any of the inclusion criteria.
* Esophageal pathology, including gastroesophageal reflux or dysphagia. Given the high frequency of presenting any of these two lasts, tests were given to the candidates to discard their presence. Two questionnaires were employed: "GERD-Q" (GastroEsophageal Disease- Questionnaire) and "EAT-10" (Eating Assesment Tool) for dysphagia.

Ages: 35 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Candidates for the study were those patients who, being planned for general surgery between January of 2017 and july of 2019, met all inclusion criteria and none of exclusion criteria. Employing a table of random numbers, patients were distributed randomly in 3 groups depending on the hypnotics they were receiving for induction of general anesthesia: propofol, etomidate or thiopental.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2017-01-10; Primary Completion 2019-07-18 (Actual); Study Completion 2019-07-18 (Actual)

PRIMARY OUTCOMES:
Change from baseline upper esophageal sphincter pressure at loss of conciousness. | Time frame: 1 minute after inserting the manometric probe, a basal measure was noted. An average of 1 minute after the hypnotic was given, once entropy had fallen below 60 or otherwise clinical signs showed unconsciousness, another measure was noted.
  Solid state high resolution manometry (Sierra Scientific Instruments, Given Imaging, Los Angeles, California Medtronic, Ireland) was used. High resolution manometry module Manoscan™ permits adquisition and recording of manometry studies. Manometric probe has a diameter of 4.2 mm and consists of 36 circunferential sensors at 1 cm intervals (Medtronic, Irlanda). Each sensor consists of 12 segments distributed radially, detecting pressures in 2.5 mm length. A pressure image is created using 432 measurement points. Sectorial pressures are averaged inside of each sensor through pressure transduction technology "Tact Array". Data adquired using manometry are represented in real time as "topographic" plots. Contour plots show different colours, each of them correspondent to a concrete pressure. Location is represented in the vertical axis and time in the horizontal axis. Data obtained using Manoscan are recorded and posteriorly analized through Manoview Software V. 3.01 (Medtronic Irlanda).

SECONDARY OUTCOMES:
Spectral Entropy | Although entropy, as all the variables, was measured through all the study, two time points were relevant: Basal and an average of 1 minuteafter the hypnotic was given. Especially important if the second measurement reached a value of 60 or less.
  Spectral entropy analyzes electroencephalographic signal and, after processing it, provides a number from 0 to 100 which is related to the level of consciousness. A patient under general anesthesia should not be over a value of 60. A sensor composed of three electrodes is placed on the forehead taking into account the electrode numbered 1 has to be located in the middle line and electrode numbered three in the temporal region avoiding the artery of the same name to prevent artefacts. Next, sensor is connected through a cable to spectral entropy monitoring module (Healthcare Technologies ®) integrated in Datex Ohmeda anesthesia machine which has been used in this study.

OTHER OUTCOMES:
upper esophageal sphincter length | 1 minute after inserting the manometric probe, a basal measure was noted. An average of 1 minute after the hypnotic was given, once entropy had fallen below 60 or otherwise clinical signs showed unconsciousness, another measure was noted.
  Employing solid state high resolution manometry not only upper esophageal sphincter pressure can be measured but also other characteristics of the sphincter such as its length. This parameter has been associated with its pressure. A high resolution manometry tool named "smart mouse" was of special usefulness to measure reliable sphincter length.
Heart rate | heart rate was monitored continuously throughout the whole study to assess the trend of its values related to two time points: basal and an average of 1 minute after the hypnotic was given.
  Continue 5 leads electrocardiogram (RA- Right Arm-, LA- Left Arm-, LL - Left Leg-, RL- Right Leg- and N- neutral-) that permit peripheral (I, II and III), unipolar (aVR- augmented vector Right-, aVL- augmented Vector Left- and aVF- augmented Vector Foot) and precordial (V1- V6) leads registry was employed. Monitor showed continuously leads II and V5 tracing; as well as computerized analysis of ST segment variation regarding isoelectric line. Also, arrhythmias analysis was kept active. Continuous electrocardiogram monitoring were carried out through General Electric hemodynamic monitoring module for S/5Avance®.
Pulse oximetry | Pulse oxymetry was monitored continuously throughout the whole study to assess the trend of its values related to two time points: basal and an average of 1 minute after the hypnotic was given.
  Its sensor was located on the opposite hand to the side were non- invasive blood pressure was measured, to avoid artefacts and interruption of registry. It was connected to the General Electric hemodynamic monitoring module for S/5Avance®. Under a value under 93% registry was interrupted.
Blood pressure | blood pressure was monitored continuously throughout the whole study to assess the trend of its values related to two time points: basal and an average of 1 minute after the hypnotic was given.
  Non invasive blood pressure monitoring was carried out through General Electric hemodynamic monitoring module for S/5Avance®. Blood pressure cuff should have the adequate length for each patient´s arm and was placed in the opposite arm where the hypnotic was given to avoid interferences with its administration. A change of heart rate or blood pressure of 20% of more over basal value was considered relevant.

CONTACTS AND LOCATIONS:
Overall Officials: Elena Sanz-Sanjosé, MD, Principal Investigator

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sivarao DV, Goyal RK. Functional anatomy and physiology of the upper esophageal sphincter. Am J Med. 2000 Mar 6;108 Suppl 4a:27S-37S. doi: 10.1016/s0002-9343(99)00337-x. PMID 10718448
- [Background] Meyer JP, Jones CA, Walczak CC, McCulloch TM. Three-dimensional manometry of the upper esophageal sphincter in swallowing and nonswallowing tasks. Laryngoscope. 2016 Nov;126(11):2539-2545. doi: 10.1002/lary.25957. Epub 2016 Mar 18. PMID 26990011
- [Background] Mei L, Dua A, Kern M, Gao S, Edeani F, Dua K, Wilson A, Lynch S, Sanvanson P, Shaker R. Older Age Reduces Upper Esophageal Sphincter and Esophageal Body Responses to Simulated Slow and Ultraslow Reflux Events and Post-Reflux Residue. Gastroenterology. 2018 Sep;155(3):760-770.e1. doi: 10.1053/j.gastro.2018.05.036. Epub 2018 May 24. PMID 29803837
- [Background] Sundman E, Witt H, Sandin R, Kuylenstierna R, Boden K, Ekberg O, Eriksson LI. Pharyngeal function and airway protection during subhypnotic concentrations of propofol, isoflurane, and sevoflurane: volunteers examined by pharyngeal videoradiography and simultaneous manometry. Anesthesiology. 2001 Nov;95(5):1125-32. doi: 10.1097/00000542-200111000-00016. PMID 11684981
- [Background] Vanner RG, Pryle BJ, O'Dwyer JP, Reynolds F. Upper oesophageal sphincter pressure and the intravenous induction of anaesthesia. Anaesthesia. 1992 May;47(5):371-5. doi: 10.1111/j.1365-2044.1992.tb02215.x. PMID 1599058
- [Background] Vanner RG, Pryle BJ, O'Dwyer JP, Reynolds F. Upper oesophageal sphincter pressure during inhalational anaesthesia. Anaesthesia. 1992 Nov;47(11):950-4. doi: 10.1111/j.1365-2044.1992.tb03196.x. PMID 1466434
- [Background] de Leon A, Ahlstrand R, Thorn SE, Wattwil M. Effects of propofol on oesophageal sphincters: a study on young and elderly volunteers using high-resolution solid-state manometry. Eur J Anaesthesiol. 2011 Apr;28(4):273-8. doi: 10.1097/EJA.0b013e3283413211. PMID 21119519
- [Background] Thorn K, Thorn SE, Wattwil M. The effects on the lower esophageal sphincter of sevoflurane induction and increased intra-abdominal pressure during laparoscopy. Acta Anaesthesiol Scand. 2006 Sep;50(8):978-81. doi: 10.1111/j.1399-6576.2006.01069.x. PMID 16923093
- [Background] Thorn K, Thorn SE, Wattwil M. The effects of cricoid pressure, remifentanil, and propofol on esophageal motility and the lower esophageal sphincter. Anesth Analg. 2005 Apr;100(4):1200-1203. doi: 10.1213/01.ANE.0000147508.31879.38. PMID 15781546
- [Background] Vakkuri A, Yli-Hankala A, Talja P, Mustola S, Tolvanen-Laakso H, Sampson T, Viertio-Oja H. Time-frequency balanced spectral entropy as a measure of anesthetic drug effect in central nervous system during sevoflurane, propofol, and thiopental anesthesia. Acta Anaesthesiol Scand. 2004 Feb;48(2):145-53. doi: 10.1111/j.0001-5172.2004.00323.x. PMID 14995935

DOCUMENTS (1):
  • Informed Consent Form (2017-01-01): https://cdn.clinicaltrials.gov/large-docs/22/NCT04413422/ICF_000.pdf